CLINICAL TRIAL: NCT04128215
Title: Sex Differences in Chronic and Acute Vascular Responses to Aerobic Exercise in Older Adults
Brief Title: Sex Differences in Vascular Responses to Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201902165- N; R21AG063143 (NIH)
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Aging
Keywords: High-Intensity Interval Training; Aerobic exercise; Acute exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Older Men (Active Comparator)
  Interventions: Behavioral: Control Period; Behavioral: Exercise Period
- Older Postmenopausal Women (Active Comparator)
  Interventions: Behavioral: Control Period; Behavioral: Exercise Period

INTERVENTIONS:
Behavioral: Control Period — Participants completed an 8-week control period of normal lifestyle.
Behavioral: Exercise Period — Participants completed an 8-week exercise intervention period of remotely supervised home-based non-weight-bearing all-extremity high intensity interval training (NWA-HIIT). NWA-HIIT consisted of 4x4-min bouts at 90% of maximal heart rate (HRmax) interspersed by 3x3-min bouts at 70% of HRmax. A 10-min warm-up and 5-minute cool-down at 70% of HRmax were included.

SUMMARY:
A key early event in cardiovascular disease development is endothelial dysfunction, characterized by impaired flow-mediated dilation. Regular aerobic exercise ameliorates endothelial dysfunction in healthy older men, but the data in healthy postmenopausal women are inconsistent with many studies showing no effect. The primary objective of this study was to examine sex differences in acute and chronic endothelial responses to exercise training in older men vs. older postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* adults able to give consent
* men and women
* women must be postmenopausal (either natural or surgical)
* 60 to 79 years of age

Exclusion Criteria:

* any relevant cardiovascular diseases (e.g., history of coronary artery bypass surgery or angioplasty, or heart failure, myocardial infarction, angina pectoris, peripheral arterial disease)
* myocardial ischemia during maximal graded exercise test
* major chronic clinical disease (e.g., diabetes, renal or hepatic disease or infection with hepatitis B, C, or HIV)
* seizures, or other relevant on-going or recurrent illness
* recent (within 3 months) or recurrent hospitalizations
* systolic blood pressure < 100 mmHg
* body mass index > 35 kg/m^2
* >5% weight change in past 3 months or unwilling to remain weight stable during study participation
* use of tobacco products including smoking traditional or e-cigarettes
* use of hormone replacement therapy in women or men (e.g., estrogen, progesterone or testosterone)
* regular aerobic exercise training (≥30 min/session and ≥ 3 days/week)

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Demetra Christou, PhD, Principal Investigator — University of Florida
Locations (1):
- Integrative Cardiovasculal Physiology Laboratory, University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Older Men; Older Postmenopausal Women: Control Period: Subjects will complete an 8-week control period of normal lifestyle, followed by the 8-week exercise period.
  Exercise Period: Subjects will complete an 8-week non-weight-bearing all-extremity high intensity interval training (NWA-HIIT). NWA-HIIT will consist of 4x4-min bouts at 90% of maximal heart rate (HRmax) interspersed by 3x3-min bouts at 70% of HRmax. A 10-min warm-up and 5-minute cool-down at 70% of HRmax will be included.
Period: Overall Study
Arm/Group | Older Men | Older Postmenopausal Women
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Older Men | Older Postmenopausal Women | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 3 | 8 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (6) | 68 (5) | 68 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 11 | 11
  Male | 9 | 0 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 11 | 20
Flow Mediated Dilation [Mean (Standard Deviation); unit: % of flow mediated dilation] | 3.41 (0.89) | 3.38 (1.73) | 3.39 (1.38)

OUTCOME MEASURES:

1. Primary Outcome: Change in FMD in Response to Chronic HIIT
Description: Flow mediated dilation (FMD) is an established non-invasive measure of endothelial function. Brachial artery FMD was determined via ultrasonography in response to reactive hyperemia following 5-min forearm ischemia. FMD was expressed as % change and was calculated as (max diameter-baseline-diameter)/baseline diameter)*100. The change in FMD for the control period was calculated as the difference in FMD from baseline to the end of the 8-week control period. The change in FMD for the exercise intervention period was calculated as the difference in FMD from the end of the 8-week control period to the end of the 8-week intervention period.
Time Frame: From baseline to end of 8-week control period; From end of 8-week control period to end of 8-week exercise intervention
Measure: Mean (Standard Deviation); unit: % flow mediated dilation
Arm/Group | Older Postmenopausal Women | Older Men
Number analyzed (Participants) | 11 | 9
% flow mediated dilation
  Control period | 0.11 (1.27) | 0.57 (2.07)
  Exercise intervention | 0.81 (1.78) | 0.10 (2.36)

2. Primary Outcome: Change in FMD in Response to Acute HIIT in the Untrained State
Description: Flow mediated dilation (FMD) is an established non-invasive measure of endothelial function. Brachial artery FMD was determined via ultrasonography in response to reactive hyperemia following 5-min forearm ischemia. FMD was expressed as % change and was calculated as (max diameter-baseline-diameter)/baseline diameter)*100. FMD was investigated at pre-exercise, at the end of a HIIT session, and 1-hour and 24-hours following a HIIT session in the untrained state (before beginning the 8-week exercise intervention consisting of HIIT). The change in FMD in response to acute HIIT was calculated 1) at the end of exercise (as the difference from pre-exercise to end of exercise); 2) 1-hour post-exercise (as the difference from pre-exercise to 1-hour post-exercise) and 3) 24-hours post-exercise (as the difference from pre-exercise to 24-hours post-exercise).
Time Frame: From pre-exercise to end of exercise; From pre-exercise to 1-hour post-exercise; From pre-exercise to 24-hours post-exercise
Measure: Mean (Standard Deviation); unit: % flow mediated dilation
Groups:
- Older Men; Older Postmenopausal Women: FMD at pre-exercise, end of exercise and 1-hour and 24-hours post-exercise.
Arm/Group | Older Men | Older Postmenopausal Women
Number analyzed (Participants) | 9 | 11
% flow mediated dilation
  End of exercise | -0.46 (2.04) | 0.19 (1.85)
  1-hour post-exercise | -0.64 (1.97) | -1.28 (1.69)
  24-hours post-exercise | -0.53 (1.18) | 0.12 (1.93)

3. Primary Outcome: Change in FMD in Response to Acute HIIT in the Trained State
Description: Flow mediated dilation (FMD) is an established non-invasive measure of endothelial function. Brachial artery FMD was determined via ultrasonography in response to reactive hyperemia following 5-min forearm ischemia. FMD was expressed as % change and was calculated as (max diameter-baseline-diameter)/baseline diameter)*100. FMD was investigated at pre-exercise, at the end of a HIIT session, and 1-hour and 24-hours following a HIIT session in the trained state (at the end of the 8-week exercise intervention consisting of HIIT). The change in FMD in response to acute HIIT was calculated 1) at the end of exercise (as the difference from pre-exercise to end of exercise); 2) 1-hour post-exercise (as the difference from pre-exercise to 1-hour post-exercise) and 3) 24-hours post-exercise (as the difference from pre-exercise to 24-hours post-exercise).
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: % flow mediated dilation
Arm/Group | Older Men | Older Postmenopausal Women
Number analyzed (Participants) | 9 | 11
% flow mediated dilation
  End of exercise | 0.77 (2.24) | -0.07 (2.32)
  1-hour post-exercise | -0.66 (2.59) | -0.63 (2.15)
  24-hours post-exercise | -0.45 (1.71) | 1.35 (1.79)

4. Primary Outcome: Correlation Coefficient for the Relationship Between Acute and Chronic FMD Response to HIIT
Time Frame: Acute FMD response at 1) pre-exercise vs. end of exercise; 2) pre-exercise vs. 1-hour post-exercise; and 3) pre-exercise vs. 24-hours post-exercise. Chronic FMD response at baseline vs. end of 8-week. exercise intervention
Measure: Number; unit: Correlation coefficient
Groups:
- Older Men; Older Postmenopausal Women: Correlation coefficients of the relationship between the change in FMD from baseline to end of 8-weeks of HIIT and the change in FMD from pre-exercise to end of exercise, 1-hour and 24-hours post-exercise.
Arm/Group | Older Men | Older Postmenopausal Women
Number analyzed (Participants) | 9 | 11
Correlation coefficient
  End of exercise | -0.32 | -0.26
  1-hour post-exercise | 0 | -0.20
  24-hour post-exercise | -0.17 | 0.07

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from study enrollment through study completion, an average of 24 weeks.
Arm/Group | Older Men | Older Postmenopausal Women
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 3/9 | 8/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Older Men (N=9) | Older Postmenopausal Women (N=11)
Vomiting, dizziness (General disorders) | 0 (0) | 1 (1)
Skin allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Ecchymosis (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Arterial spasm (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT04128215/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT04128215/ICF_001.pdf